CLINICAL TRIAL: NCT01464840
Title: The Pharmacokinetics of Azithromycin Prophylaxis for Cesarean Delivery
Acronym: PKAZ
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amelia Sutton, MD, PhD, Fellow/Instructor, Maternal Fetal Medicine, University of Alabama at Birmingham
Other Study IDs: F101111007
Record Dates: First submitted 2011-10-26; First posted 2011-11-04 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Endometritis
Keywords: Pregnancy; Cesarean section; Antibiotic
MeSH Terms: conditions — Endometritis | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood, maternal adipose tissue, maternal myometrium, maternal breast milk, amniotic fluid, and fetal cord blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 15 minutes: 500 mg of intravenous azithromycin will be administered 15 minutes prior to incision.
  Interventions: Drug: Azithromycin
- 30 minutes: 500 mg of intravenous azithromycin will be administered 30 minutes prior to incision.
  Interventions: Drug: Azithromycin
- 60 minutes: 500 mg of intravenous azithromycin will be administered 60 minutes prior to incision.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 500 mg intravenous infused over 1 hour
  Other Names: Zmax

SUMMARY:
PKAZ is a single institution study designed to evaluate the optimal dosing parameters for azithromycin for pre-surgical cesarean prophylaxis.

Hypothesis: Pre-operative administration of azithromycin results in maternal and neonatal tissue concentrations that adequately treat microbes commonly involved in post-cesarean infections.

ELIGIBILITY:
Inclusion Criteria:

* Women 19 years and older
* Term (37 weeks and greater)
* Singleton gestation
* Scheduled cesarean section
* Non-laboring
* Intact membranes

Exclusion Criteria:

* < 19 years of age
* Preterm (< 37 weeks)
* Multifetal gestation
* Laboring or ruptured membranes
* Known fetal anomaly
* Oligo- or polyhydramnios
* Macrolide allergy
* Macrolide exposure within 2 weeks
* Medical co-morbidities
* Hepatic or renal impairment
* Taking medications that prolong the QT interval
* Currently taking nelfinavir, efavirenz, or flucanozole
* Structural heart defects or arrythmia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women 19 years and older undergoing scheduled cesearean sections
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amelia L Sutton, M.D., Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the prenatal clinic from May 2012 to May 2013.
Groups:
- 15 Minutes: 500 mg of intravenous azithromycin will be administered 15 minutes prior to incision.
  Azithromycin : 500 mg intravenous infused over 1 hour
- 30 Minutes: 500 mg of intravenous azithromycin will be administered 30 minutes prior to incision.
  Azithromycin : 500 mg intravenous infused over 1 hour
- 60 Minutes: 500 mg of intravenous azithromycin will be administered 60 minutes prior to incision.
  Azithromycin : 500 mg intravenous infused over 1 hour
Period: Overall Study
Arm/Group | 15 Minutes | 30 Minutes | 60 Minutes
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15 Minutes | 30 Minutes | 60 Minutes | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (4) | 27 (5) | 29 (6) | 28 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Group That Attain an Adequate Azithromycin Concentration
Description: The primary outcome of this study will be the number of patients in each group that attain an azithromycin concentration in the various maternal and fetal tissues at least equivalent to the MIC 90 for common organisms involved in post-cesarean infections.
Time Frame: 48 hours after delivery
Population: No patients had azithromycin concentrations at least equivalent to the MIC 90.
Measure: Number; unit: number of participants
Arm/Group | 30 Minutes | 15 Minutes | 60 Minutes
Number analyzed (Participants) | 10 | 10 | 10
number of participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 15 Minutes | 30 Minutes | 60 Minutes
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No